CLINICAL TRIAL: NCT03132779
Title: Intralipid Related Effect on NKcells in Patients With Unexplained Recurrent Spontaneous Abortions
Brief Title: Intralipid Related Effect on NKcells in Patients With Unexplained Recurrent Spontaneous Abortion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Mohamed Bahaa Eldin Ahmed (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, Clinical professor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intralipid
Record Dates: First submitted 2017-04-16; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Miscarriage
Keywords: Intralipid; NK cells; Recurrent miscarriage
MeSH Terms: conditions — Abortion, Habitual | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Intervention Model Description: Women with unexplained recurrent spontaneous abortions having increased NKcells activity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One armed (Experimental): One group of patient will take Intralipid for all
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Intralipid — Adose of intralipid given and rechecking NKcells activity
  Other Names: Intralipid 18 mg

SUMMARY:
Evaluating the effect of intralipid on the natural killer cells

DETAILED DESCRIPTION:
This study will done on women with recurrent spontaneous abortions having increased NKCELLS activity and evaluate the effect of Intralipid on them after re-estimation of NKcells activity again after one week of Intralipid adminstration

ELIGIBILITY:
Inclusion Criteria:

* All women icluded having recurrent spontaneous abortions equal or more than twice.
* Alittle women having increased NKCELLS activity.

Exclusion Criteria:

* Any other diseases causing miscarriage as autoimmune (lupus erythematosus or antiphospholipid antibodies syndrome )or endocrinopathy (diabetes mellitus, thyroid disorders and hyperprolactinaemia)or thrombophilia (factor v leiden mutation, protein c or s deficiency, prothrombin G20210A mutation, antithrombin III deficiency ) or abnormal karyotyping to one or both of parents or previous history of hormonal contraception or intrauterine device usage at last 3 months or any contraindications for intralipid usage.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with recurrent spontaneous abortions
Enrollment: 34 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-01-20 (Estimated); Study Completion 2018-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in NK cells activity after injection of intralipid | One week
  NK cells is measured before and after injection of intralipid and is noticed for change in activity

CONTACTS AND LOCATIONS:
Overall Officials: Hassan T Khairy, Professor, Study Director — Hassan Tawfik office

IPD SHARING:
Plan to Share IPD: Undecided